CLINICAL TRIAL: NCT04499898
Title: Randomized Controlled Trial of Carvedilol Versus Endoscopic Band Ligation for Primary Prophylaxis of Oesophageal Variceal Bleeding in Cirrhotic Patients With Arterial Hypertension
Brief Title: Carvedilol Versus Endoscopic Band Ligation for Primary Prophylaxis of Oesophageal Variceal Bleeding
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: nabeela protocol
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carvedilol (Experimental): Carvedilol
  Interventions: Drug: Carvedilol
- Band Ligation (Active Comparator): Band Ligation
  Interventions: Procedure: Endoscopic band ligation

INTERVENTIONS:
Drug: Carvedilol — Carvedilol
  Other Names: carvid
  Arms: carvedilol
Procedure: Endoscopic band ligation — Endoscopic band ligation
  Other Names: band ligation
  Arms: Band Ligation

SUMMARY:
Carvedilol versus endoscopic band ligation for primary prophylaxis of oesophageal variceal bleeding in cirrhotic patients with arterial hypertension

DETAILED DESCRIPTION:
A Randomized controlled trial of carvedilol versus endoscopic band ligation for primary prophylaxis of oesophageal variceal bleeding in cirrhotic patients with arterial hypertension

ELIGIBILITY:
Inclusion Criteria:

* • Aged >18 years

  * Cirrhotic patients with arterial hypertension
  * Endoscopic evidence of medium/large-sized esophageal varices

Exclusion Criteria:

* • History of variceal bleeding or previous primary prevention of varices.

  * Portal vein thrombosis or previous porto-systemic shunts as TIPS.
  * Patients on drugs affecting portal pressure (beta blockers, nitrates).
  * Advanced cardiovascular disease including acute myocardial infarction, atrio-ventricular block, congestive heart failure, chronic peripheral ischemia, severe bradycardia.
  * Patients with severe respiratory diseases (COPD, bronchial asthma).
  * Uncontrolled diabetes mellitus
  * Renal impairment
  * Hepatocellular carcinoma
  * Allergy to carvedilol
  * Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with the first variceal bleeding within 1 year | 1 year
  The number of patients with the first variceal bleeding within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, Prof, Study Director — Tanta University - Faculty of Medicine; Nabila Abd El-Nasser Abd El-Wahed El-Gazzar, ass. lect, Principal Investigator — Tanta University Faculty of medicine
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No